CLINICAL TRIAL: NCT03778021
Title: Engaging Navajo Elementary Schools in Randomized Controlled Trial of Yeego! Healthy Eating & Gardening
Brief Title: Yeego! Healthy Eating & Gardening School-Based Randomized Controlled Trial
Acronym: Yeego!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shirley Beresford, Professor, Cancer Prevention Program, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RG1001953; 8716 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2018-03752 (Registry Identifier: NCI / CTRP); U54CA132381-11 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-11

CONDITIONS: Dietary Habits; Health Behavior; Eating Behavior
MeSH Terms: conditions — Feeding Behavior; Health Behavior | interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Group Randomized Trial
Who Masked: Outcomes Assessor
Masking Description: Interviewers were not informed of school or school assignment at follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention schools receive a raised bed school garden and a curriculum of healthy eating and gardening lessons.
  3rd and 4th grade students in the intervention group received the curriculum and exposure to the school garden during the academic school year (2019-20)
  Behavioral Gardening Exposure: Assistance provided with planting and maintaining the school garden
  Healthy Eating and Gardening Curriculum: 14 to 17 lessons (about 45 minutes each) throughout the school year, during the normal school day, that are focused on healthy eating and gardening, coordinated with the growing season.
  Interventions: Behavioral: Behavioral Gardening Exposure; Behavioral: Healthy Eating and Gardening Curriculum
- Comparison Group (No Intervention): For the comparison group schools, no program was provided in school year (2019-2020).
  After the trial, and the follow-up evaluation, in school year 2020-2021 comparison schools received delayed intervention components as follows: School gardens were created during the 2020-2021 school year (subject to delays due to pandemic restrictions). Curriculum materials were supplied to the school for use by teachers as they saw fit, after pandemic restrictions were lifted.

INTERVENTIONS:
Behavioral: Behavioral Gardening Exposure — Assistance provided with planting and maintaining the school garden
  Arms: Intervention Group
Behavioral: Healthy Eating and Gardening Curriculum — 14 to 17 lessons (about 45 minutes each) throughout the school year, during the normal school day, that are focused on healthy eating and gardening, coordinated with the growing season
  Arms: Intervention Group

SUMMARY:
In this study, one year changes in healthy eating and gardening behaviors associated with the intervention were estimated using a group randomized controlled trial design, with the comparison arm receiving a delayed intervention in the following school year.

DETAILED DESCRIPTION:
The small randomized controlled trial of an intensive curriculum and school garden intervention was implemented in elementary schools in two communities (Shiprock and Tsaile). The study began in year 1 with a period of engagement and recruitment of schools in each community; with the goal of recruiting three schools in each community to complete the run-in phase. The run-in period included time for greater engagement with the school community, an assessment of the potential garden site and an assessment of evaluation readiness. Depending on whether three schools in the community qualify for the study at the end of run-in, or only two schools per community, it was planned to randomize three or two schools to intervention or delayed intervention status in each community. Six schools were randomized, two intervention schools and 4 comparison (delayed intervention) schools. Baseline data collection was conducted at the beginning of the school year 2019-2020 in Year 2 with 3rd and 4th grade children. Students in the intervention schools received the curriculum and school garden during that academic school year (Study Year 2). At the end of the school year, 8-month follow-up assessment was conducted. The main evaluation period is between baseline and 8-month follow-up, and the statistical analysis methods estimate the differential change in outcome measures (healthy eating and gardening).

Not part of the clinical trial, the study continued in the next school year (2020-2021). At the beginning of Study Year 3, the comparison schools were scheduled to receive the delayed intervention. During Study Year 3, it was planned to conduct quarterly community gardening workshops for adult family members in all schools. Due to the COVID-19 pandemic, a series of 10 video workshops were produced and made available via YouTube. Attendance/Views were tracked. A final assessment survey was conducted at the end of that school year (in 2021) in all 6 schools to allow additional descriptive analyses.

ELIGIBILITY:
Inclusion Criteria:

* Elementary schools in Tsaile and Shiprock will have been in existence for at least three years, school size (have between 40 to 100 students in grades 3 and 4 combined), have more than two-thirds Navajo students and satisfy a garden site checklist that can overcome garden barriers (e.g. have access to water)
* Assessment is restricted to Male/female students in grades 3 and 4 attending school in either Tsaile or Shiprock

Exclusion criteria:

* Students in grades other than 3rd or 4th are not eligible for assessment

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 294 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Beresford, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Agricultural Science Center at Farmington, College of Agricultural, Consumer, and Environmental Sciences, New Mexico State University, Farmington, New Mexico
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lombard KA, Beresford SAA, Ornelas IJ, Jim J, Bauer M, Nez F. Where health and horticulture intersect: A Navajo wellness collaboration. HortScience. 2015;50(9):S360.
- [Background] Lombard KA, Beresford SA, Ornelas IJ, Topaha C, Becenti T, Thomas D, Vela JG. Healthy gardens/healthy lives: Navajo perceptions of growing food locally to prevent diabetes and cancer. Health Promot Pract. 2014 Mar;15(2):223-31. doi: 10.1177/1524839913492328. Epub 2013 Jul 12. PMID 23855020
- [Background] Lombard KA, Forster-Cox S, Smeal D, O'Neill MK. Diabetes on the Navajo nation: what role can gardening and agriculture extension play to reduce it? Rural Remote Health. 2006 Oct-Dec;6(4):640. Epub 2006 Oct 16. PMID 17044752
- [Background] Ornelas IJ, Deschenie D, Jim J, Bishop S, Lombard K, Beresford SA. Yeego Gardening! A Community Garden Intervention to Promote Health on the Navajo Nation. Prog Community Health Partnersh. 2017;11(4):417-425. doi: 10.1353/cpr.2017.0049. PMID 29332855
- [Background] Ornelas IJ, Rudd K, Bishop S, Deschenie D, Brown E, Lombard K, Beresford SAA. Engaging School and Family in Navajo Gardening for Health: Development of the Yeego Intervention to Promote Healthy Eating among Navajo Children. Health Behav Policy Rev. 2021 May;8(3):212-222. doi: 10.14485/HBPR.8.3.3. Epub 2021 May 1. PMID 34901297
- [Result] Beresford SAA, Ornelas IJ, Bauer MC, Garrity GA, Bishop SK, Francis B, Rillamas-Sun E, Garcia LV, Vecenti FSA, Lombard KA. Group Randomized Trial of Healthy Eating and Gardening Intervention in Navajo Elementary Schools (Yeego!). AJPM Focus. 2022 Sep 16;1(2):100033. doi: 10.1016/j.focus.2022.100033. eCollection 2022 Dec. PMID 37791240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two areas of the Navajo Nation were selected. Elementary schools within 70 miles of the closest Diné College campus were identified.
  Eligibility criteria for schools included within 30 miles of one of the two campuses; number of 3rd and 4th grade students between 40 and 140.
  Ten schools were eligible for recruitment. 6 schools completed run-in.
Pre-assignment Details: Recruitment-eligible schools were 5 in each area. These schools were listed in random order within area. 9 schools started run-in, one school was not contacted. Two schools failed run-in, one in each area, leaving 6 schools eligible to be randomized.
  In 2019, six schools completed run-in and were randomized to intervention (2) or delayed intervention (4).
Units Other Than Participants: Schools
Groups:
- Intervention Group: Intervention schools receive a raised bed school garden and a curriculum of healthy eating and gardening lessons.
  3rd and 4th grade students in the intervention group received the curriculum and exposure to school garden during the academic school year (2019-20)
  Behavioral Gardening Exposure: Assistance provided with planting and maintaining the school garden
  Healthy Eating and Gardening Curriculum: 14 to 17 lessons (about 45 minutes each) throughout the school year, during the normal school day, that are focused on healthy eating and gardening, coordinated with the growing season.
- Comparison Group: For the comparison group schools, no program was provided in school year (2019-2020).
  After the trial, and the follow-up evaluation, comparison schools received delayed intervention components as follows: School gardens were created during the 2020-2021 school year (subject to delays due to pandemic restrictions). Curriculum materials were supplied to the school for use by teachers as they saw fit, after pandemic restrictions were lifted.
Period: Overall Study
Arm/Group | Intervention Group | Comparison Group
Started (Schools were the unit of randomization. School was the unit of intervention. Evaluation used data from students in each participating school. Details about baseline characteristics and results of evaluation all rely on student data.) | 100; 2 Schools | 194; 4 Schools
Completed (At the student level, completion refers to providing follow-up data. At the school level, completion refers to completion of intervention or comparison condition, and of permission to collect follow up data from the students. All students in grade 3 or 4 in the schools were exposed to the intervention condition to which their school was assigned.) | 72; 2 Schools | 141; 4 Schools
Not Completed | 28; 0 Schools | 53; 0 Schools
Not completed — Student failed to respond to follow-up survey | 28 | 53

BASELINE CHARACTERISTICS:
Population: School was unit of randomization, and unit of intervention delivery to 3rd and 4th grade students.
  3rd and 4th grade student participants completed baseline. Participant was the unit analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Comparison Group | Total
Number analyzed (Participants) | 100 | 194 | 294
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.6 (0.7) | 8.7 (0.9) | 8.7 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 109 | 151
  Male | 58 | 85 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 91 | 175 | 266
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 3 | 8 | 11
  Unknown or Not Reported | 1 | 8 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 194 | 294
Understands Navajo [Count of Participants; unit: Participants] | 49 | 119 | 168
BMI for age percentile [Mean (Standard Deviation); unit: percentile] | 73.1 (31.2) | 69.7 (29.8) | 70.9 (30.3)
Overweight or Obese [Count of Participants; unit: Participants] — Percent overweight or obese (%)
  Participants | 50 | 83 | 133
Self-efficacy to eat F&V [Mean (Standard Deviation); unit: units on a scale] — Self-efficacy to eat Fruits and Vegetables (F&V) is a scale made up of the average of five items each with four-point Likert scale responses (I know I can, I think I can, I'm not sure I can, and I know I can't). Score range is 1 to 4. Higher scores represents higher self-efficacy.
  units on a scale | 3.2 (0.65) | 3.4 (0.57) | 3.3 (0.60)
AHEI Healthy Foods Score [Mean (Standard Deviation); unit: units on a scale] — The Healthy Foods Score is a subscale from the modified Alternative Healthy Eating Index (AHEI). Data for the modified AHEI were derived from a picture sort frequency tool, estimating frequencies of consumption of ten major food groups of the Navajo diet. Scoring published as AHEI-2010 was applied.
  The subscale, the Healthy Foods Score, is the sum of scores for fruits (fresh & dried), vegetables (not salad), whole grains, beans, nuts, only. The minimum value is 0 and the maximum is 36. Higher values represent a better outcome.
  .
  units on a scale | 16.9 (5.8) | 17.8 (6.4) | 17.5 (6.2)
Full self-efficacy to grow F&V at school [Number; unit: percentage of participants] — Percent of participants reporting "I know I can". This binary variable was derived from a question about student's confidence to grow F&V at school. The question had responses on a 4-point Likert scale. Only the "I know I can" point was used to create the binary variable for full self-efficacy to grow F&V at school.
  percentage of participants | 49.0 | 40.0 | 43.2

OUTCOME MEASURES:

1. Primary Outcome: Estimated Change in Child Fruit & Vegetable Self-efficacy
Description: Self-efficacy for eating F&V score is average of responses to five 4-point Likert scale questions. Higher score is higher self-efficacy. Score range is 1 to 4.
  Change in self-efficacy is based on a model that uses all available data (from baseline and 8-month follow-up). The unit of analysis is participant-timepoint. The analysis accounts for nesting within schools.
  Using a repeated measures linear mixed model analysis, the results are estimated change in self-efficacy score from baseline to 8-month follow-up, contrasting intervention group to comparison group.
  From the model, the estimated change in scores from baseline to 8-month follow-up ranged from 0.14 to 0.62. The unit of measure is "score on a scale". The results show the least squares estimate of change in that score.
  Positive estimated change in score indicates self-efficacy increased from baseline to follow-up.
  Positive differential change indicates that intervention group change was greater than comparison group.
Time Frame: Beginning to end of school year 2019-20 ( Baseline and ~ 8 months)
Population: Participants were 3rd and 4th grade students responding to baseline and/or 8-month follow-up. The participant at specified time point was the unit of analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: participant-time point
Arm/Group | Intervention Group | Comparison Group
Number analyzed (Participants) | 100 | 194
Number analyzed (participant-time point) | 172 | 335
score on a scale | 0.47 (0.08) | 0.24 (0.05)
Statistical Analysis 1: Comparison: Intervention Group vs Comparison Group; The unit of measure is "score on a scale". The results show the least squares estimate of change in that score, from baseline to 8-month follow-up in each group from model. Values from the 100 and 194 baseline respondents and from the 72 and 141 follow-up respondents of intervention and comparison groups respectively contributed to the repeated measures linear mixed model, where the units of analysis were participant-time. The nesting within schools was accounted for in the model; Test type: Superiority; p = 0.017, Mixed Models Analysis — Estimated differential change in score between intervention and comparison group from repeated measures linear mixed model. All the reported analyses conservatively specified covariance structure as general covariance (unstructured). alpha = 0.05; Repeated measures linear mixed model analysis. Student nested within school. Model fit time, intervention and time by intervention interaction; Mean Difference (Net) = 0.22, 95% CI 2-sided [0.04 to 0.41], Standard Error of Mean 0.093 — Estimated differential change (intervention minus control) from repeated measures linear mixed model; In the repeated measures linear mixed model, time was treated as a fixed effect. In the specification of the repeated measures linear mixed model, students were nested within schools. All the reported analyses conservatively specified covariance structure as general covariance (unstructured)

2. Primary Outcome: Estimated Change in AHEI Healthy Foods Score
Description: The Healthy Foods Score is a subscale from the modified Alternative Healthy Eating Index (AHEI). Data were derived from a picture sort frequency tool estimating consumption frequencies of ten major food groups of the Navajo diet. Scoring used the published AHEI-2010.
  The subscale is the sum of scores for fruits (fresh & dried), vegetables (not salad), whole grains, beans, nuts, only. Values range from 0 to 36. Higher values represent a better outcome.
  Change in Score is based on a model that uses all available data (from baseline and 8-month follow-up).
  The model is from a repeated measures linear mixed model analysis. Change in Healthy Foods score is estimated from baseline to 8-mth follow-up, contrasting intervention group to comparison group. The change scores ranged from -0.63 to 3.66.
  Positive estimated change indicates an increase from baseline to follow-up. Positive differential change indicates that intervention group change was greater than comparison group change.
Time Frame: Beginning to end of school year 2019-20 ( Baseline and ~ 8 months).
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: participant-time point
Arm/Group | Intervention Group | Comparison Group
Number analyzed (Participants) | 100 | 194
Number analyzed (participant-time point) | 172 | 335
score on a scale | 1.98 (0.85) | 0.58 (0.61)
Statistical Analysis 1: Comparison: Intervention Group vs Comparison Group; Results present estimated change in score from baseline to 8-month follow-up in each group from model. Values from the 100 and 194 baseline respondents and from the 72 and 141 follow-up respondents of intervention and comparison groups respectively contributed to the repeated measures linear mixed model, where the units of analysis were participant-time. The nesting within schools was accounted for in the model; Test type: Superiority; p = 0.18, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.41, 95% CI 2-sided [-0.66 to 3.49] — Estimated differential change from baseline to follow-up from model (intervention minus control); In the repeated measures linear mixed model, time was treated as a fixed effect. In the specification of the repeated measures linear mixed model, students were nested within schools

3. Primary Outcome: Estimated Ratio of Full Self-efficacy to Grow F&V at School
Description: Measure derived from Percent of participants at each time point reporting "I know I can".
  Using generalized mixed models, specifying a binomial distribution, accounting for nesting within schools, the Odds ratio of 8-month follow-up to baseline percent reporting "I know I can" was estimated for both intervention and comparison groups. The overall range in these odds ratios was 0.95 to 3.63 .
  The contrast of intervention group to comparison group was also an odds ratio.
Time Frame: Beginning to end of school year 2019-20 ( Baseline and ~ 8 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: odds ratio
Units Other Than Participants: participant-time point
Groups:
- Comparison Group: .For the comparison group schools, no program was provided in school year (2019-2020).
  After the trial, and the follow-up evaluation, comparison schools received delayed intervention components as follows: School gardens were created during the 2020-2021 school year (subject to delays due to pandemic restrictions). Curriculum materials were supplied to the school for use by teachers as they saw fit, after pandemic restrictions were lifted.
Arm/Group | Intervention Group | Comparison Group
Number analyzed (Participants) | 100 | 194
Number analyzed (participant-time point) | 172 | 335
odds ratio | 1.92 [1.02 to 3.63] | 1.48 [0.95 to 2.31]
Statistical Analysis 1: Comparison: Intervention Group vs Comparison Group; Odds ratio of 8-month follow-up to baseline percent reporting " I know I can" was estimated from repeated measures generalized linear mixed model with binomial distribution. Values included from the 100 and 194 baseline respondents and from the 72 and 141 8-month follow-up respondents of intervention and comparison groups respectively. The person-timepoint is the unit of analysis; Test type: Superiority; p = 0.51, Mixed Models Analysis — Repeated measures generalized linear mixed model with binomial distribution (variable was "I know I can" - yes versus no); The odds of the odds ratio is reported as the intervention effect; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.60 to 2.81] — Odds ratio from estimated least squares from generalized mixed model with binomial distribution specified. Intervention odds of change compared to comparison group odds of change via odds ratio

ADVERSE EVENTS:
Time Frame: Up to 1 year 8 months
Arm/Group | Intervention Group | Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/194
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/194
Other Adverse Events (participants affected / at risk) | 0/100 | 0/194

LIMITATIONS AND CAVEATS:
The group randomized trial was small, in that only six schools were enrolled and randomized. Not all 3rd and 4th graders participated in the baseline assessment.

Not all students completing baseline also completed follow-up. Only six of the 11 standard components of AHEI could be estimated. Dietary behaviors were assessed using self-efficacy for F&V, and metrics based on the picture sort tool. Neither of these methods is considered as reliable as the 24 hour recall.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT03778021/Prot_SAP_000.pdf